CLINICAL TRIAL: NCT05850884
Title: Evaluation of Intestinal Parasites in Patients With Intestinal Cancer in Sohag, Egypt.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Ibrahim Selim, Teaching Assistant, Sohag University
Other Study IDs: Soh-Med-23-04-24MS_
Record Dates: First submitted 2023-04-30; First posted 2023-05-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Intestinal Parasites in Patients With Intestinal Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: • One hundred stool samples will be collected from patients with intestinal cancer admitted to Sohag Hospital.
  Interventions: Diagnostic Test: stool examination
- group B: one hundred stool samples will be collected from the control group of patients who attended outpatient clinics
  Interventions: Diagnostic Test: stool examination

INTERVENTIONS:
Diagnostic Test: stool examination — Each collected sample will be divided into three parts; 1st part will be examined freshly without preservatives by macroscopic and microscopic examination, the 2nd part will be preserved for concentration techniques, staining, and microscopic examination and the 3rd part will be cultivated for Strongyloides stercoralis diagnosis

SUMMARY:
This study aims to evaluate the intestinal parasitic infections in patients with intestinal cancer in comparison to non-cancer individuals

DETAILED DESCRIPTION:
Intestinal parasitic infections continue to be characterized as a significant cause of morbidity worldwide, and according to World Health Organization (WHO) statistics, more than a quarter of the world's population, mostly in developing countries, are infected Acquisition of infection, clinical severity, and outcome of a parasitic disease depend on innate and acquired host immunity as well as on the parasite's response against the host when the infection is established Chronic infections and inflammation along with unhealthy diet, stressful lifestyle, cell damage, constant exposure to radiation, and harmful chemicals are risk factors for the development of cancers As infectious factors, the Blastocystis hominis and Cryptosporidium spp. are opportunistic protozoa isolated from the human host gastrointestinal tract, These prevalent enteric parasites may cause serious challenges in people undergoing colorectal cancer treatment (chemotherapy)

ELIGIBILITY:
Inclusion Criteria:

* intestinal cancer patients (colorectal cancer, intestinal lymphoma, gastrointestinal stromal tumors, and other malignant variants)

Exclusion Criteria:

* patient took antibiotics within the previous four weeks and anti-parasitic drugs within the previous two weeks

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Case-control study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
evaluate the intestinal parasitic infections in patients with intestinal cancer in comparison to non-cancer individuals | 12 months
  • Each collected sample will be divided into three parts; 1st part will be examined freshly without preservatives by macroscopic and microscopic examination, the 2nd part will be preserved for concentration techniques, staining, and microscopic examination and the 3rd part will be cultivated for Strongyloides stercoralis diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: nada a elnady, professor, Study Director — Sohag University; emad e nabil, ass prof, Study Chair — Sohag University; manal r gaballah, lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided